CLINICAL TRIAL: NCT02009475
Title: The Effect of Two Exercise Training Protocols on Physiological and Biochemical Parameters in Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Robert Klempfner Heart Rehabilitation Institute (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Robert Klempfner Heart Rehabilitation Institute, Director Cradiac Rehabilitation Institute, Sheba Medical Center, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LACT_HF_KIN
Record Dates: First submitted 2013-12-02; First posted 2013-12-12 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Rehabilitation; Exercise Training; Interval training
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continues aerobic training (Active Comparator): Treadmill or exercise bike training with target heart rate of 50-70% of the heart rate reserve (or 50-60% of the peak VO2 reserve). Overall 45 minutes of exercise (including the 5-10 minute warm-up period).
  Interventions: Other: Continues aerobic training
- Interval Exercse Training (Experimental): Bouts of high intensity interval treadmill or exercise bike training, comprising of 85-95% of the heart rate reserve (or 80-90% of the peak VO2 reserve), for the duration of 4 minutes, separated by periods of low intensity activity until the heart rate reaches 50% of the peak heart rate. This set will be repeated 3 times.
  Interventions: Other: Interval exercise training

INTERVENTIONS:
Other: Interval exercise training
  Arms: Interval Exercse Training
Other: Continues aerobic training
  Arms: Continues aerobic training

SUMMARY:
The aim of the present study is to evaluate differential lactate removal kinetics in heart failure patients that are trained according to 2 different exercise protocols:

(A) High intensity intervals training (HIT); (B) Continuous moderate aerobic training (MAT)

DETAILED DESCRIPTION:
Introduction: Congestive heart failure (CHF) patients suffer from early fatigue and functional aerobic impairment. Their reduced cardiac output and O2 delivery to the peripheral muscles shifts those patients consistent anaerobic metabolism, thus, CHF patients rely on anaerobic metabolism even in everyday life activity. This metabolism leads to a shift of muscles fiber types from mainly slow twitch, oxidative type I fibers to fast twitch, glycolytic type IIb fibers. Monocarboxylate proteins MCT1 and MCT4 transport lactate crosses the membrane. MCT1 is responsible for the lactate uptake and MCT4 is responsible for efflux of excess lactate. Exercise training is known to improve the quality of life in CHF. We hypothesized that exercise training might change MCT1 and 4 expression and distribution. Accordingly, these changes may also affect lactate clearance during recovery, which may contribute to the beneficial effect of exercise training in CHF patients. Methods: New-York Heart association (NYHA) class II-III CHF patients will be assigned to the experiment. At baseline and upon training conclusion they will undergo the same tests battery. The test battery includes heart rate, blood pressure measurements, echocardiographic evaluation. All participants will fill out "Minnesota living with heart failure" questionnaire. Subsequently, after their basal blood lactate will be assessed they will undergo measurement which will be followed by lactate clearance-rate evaluation.

Randomly each patient will then be assigned to one of two experimental training groups: (A) High intensity intervals training (HIT); (B) Continuous moderate aerobic training (MAT). Each volunteer will be trained twice a week for 12 weeks, according to his/hers assigned training protocol and in accordance to exercise training guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Stable heart failure patients referred to exercise training in a tertiary care cardiac rehabilitation institute
* Age > 21

Exclusion Criteria:

* Severe symptomatic heart failure
* Severe orthopedic limitations
* Unstable arrythmia
* Cognitive decline or substance abuse
* Unable to comply with exercise protocol
* Significant pulmonary disease
* NYHA 4 heart failure class

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Lactate clearance kinetics | Baseline and following 12 weeks of training
  Change from baseline of lactate clearance kinetics followoing a 12 weeks exercise program based on two different training protocol (continues and interval training)

SECONDARY OUTCOMES:
Peak VO2 change | Pre- and post 12 week exercise program
  Change from baseline of the peak VO2 following the 12 weeks exercise program

OTHER OUTCOMES:
Quality of life questioner (MLWHF) | Pre training and 12 weeks later post exercise training period

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Cardiac Rehabilitation Institute, Tel Hashomer , Ramat Gan, Israel